CLINICAL TRIAL: NCT04267952
Title: The Effect of the Theory of Planned Behaviour Based Hand Hygiene Intervention Program on Primary School Students' Health Outcomes and Absenteeism in School
Brief Title: Hand Hygiene Intervention Program on Primary School Students' Health Outcomes and Absenteeism in School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Gulcin Uyanık, Research Assistant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 509055
Record Dates: First submitted 2019-12-21; First posted 2020-02-13 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Tract; Infection, Upper (Acute); Hand Hygiene; Absenteeism
Keywords: Health education; Theory of planned behavior; Primary schools
MeSH Terms: conditions — Infections; Health Education

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participation will not know whether they are in the experimental or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first group (Experimental): Hand hygiene intervention program prepared by using planned behavior theory will be applied to the students in this group.
  Interventions: Behavioral: Hand hygiene intervention program developed according to planned behavior theory
- second group (Active Comparator): Students in this group will be given classic hand hygiene training
  Interventions: Behavioral: Classical hand hygiene education

INTERVENTIONS:
Behavioral: Hand hygiene intervention program developed according to planned behavior theory — The perception of the importance of hand hygiene with expression of damages of microorganisms (stories about illnesses etc.). Visually assisted hand hygiene training experiments to ensure the visibility of microorganisms in the environment. Demonstration and application of the correct hand washing technique with music. All applications will take place in three lessons (120-minute).
  Arms: first group
Behavioral: Classical hand hygiene education — expression of hand hygiene with verbal presentation method in a 40-minute lecture
  Arms: second group

SUMMARY:
The most common infections in schools are acute respiratory infections (colds, pharyngitis, influenza and others) and diarrheal diseases. The incidence of these infections may also be an important cause of school absenteeism, leading to negative outcomes in both education and health.

WHO states that handwashing a well-known primary infection control measure, is the most important hygiene measure to prevent the spread of infection when handwashing is done with soap and water. Since behavioral choices that determine lifestyle are made in childhood, it is important that health education in hand hygiene be implemented as early as possible to improve healthy behaviors. In this context, schools are important structures for information and behavior change about water, sanitation and hygiene interventions.

Planned Behavior Theory (PBT) states that intention is the main precursor of behavior. According to the theory, intention is guided by three independent variables (perceived behavior control, attitudes and subjective norms), and intention formation leads to the development of behavior. The theory has been used in a study to improve hand hygiene behavior in health workers, but it has not been used in the literature to improve hygiene behaviors in children.

Researches indicate that students who do not attend school frequently or for a long time have difficulty in mastering the subject described in the lesson and that school absenteeism is an issue that should be emphasized in education. Therefore, hand hygiene has a simultaneous effect that improves both education and health and contributes to a safe and healthy learning environment. The aim of this research is; To test the effect of hand hygiene intervention program based on Planned Behavior Theory on students' health outcomes and school absenteeism.

DETAILED DESCRIPTION:
The most common infections in schools are acute respiratory infections (colds, pharyngitis, influenza and others) and diarrheal diseases. Acute respiratory infections are a major cause of morbidity and mortality in children and a major public health problem in both developed and developing countries. The incidence of these infections may also be an important cause of school absenteeism, leading to negative outcomes in both education and health.

Improving water, sanitation and hygiene in schools is an important intervention for the healthy development of children. WHO states that handwashing a well-known primary infection control measure, is the most important hygiene measure to prevent the spread of infection when handwashing is done with soap and water. It was found that well-structured and applied handwashing techniques were useful in reducing the incidence of gastro-intestinal and respiratory infections in school children; handwashing with soap reduces respiratory infections in children by 16% - 25%.

In children, unlike adults, it is more likely to give positive behavior because negative hygiene habits are less established and do not have stereotyped and difficult to change habits. Since behavioral choices that determine lifestyle are made in childhood, it is important that health education in hand hygiene be implemented as early as possible to improve healthy behaviors. In this context, schools are important structures for information and behavior change about water, sanitation and hygiene interventions. Hand hygiene initiatives in the school provide multiple gains by enabling children to become hygienic ambassadors in their own homes and gaining the skills they can sustain during the adult period.

Planned Behavior Theory (PBT) states that intention is the main precursor of behavior.

According to the theory, intention is guided by three independent variables (perceived behavior control, attitudes and subjective norms), and intention formation leads to the development of behavior. In a systematic review of 30 studies using PBT in various health interventions, two thirds of studies reported effective behavior change. The theory has been used in a study to improve hand hygiene behavior in health workers, but it has not been used in the literature to improve hygiene behaviors in children.

Researches indicate that students who do not attend school frequently or for a long time have difficulty in mastering the subject described in the lesson and that school absenteeism is an issue that should be emphasized in education. Therefore, hand hygiene has a simultaneous effect that improves both education and health and contributes to a safe and healthy learning environment. The aim of this research is; To test the effect of hand hygiene intervention program based on Planned Behavior Theory on students' health outcomes and school absenteeism.

ELIGIBILITY:
Inclusion Criteria:

* primary school student (especially third and fourth class student)

Exclusion Criteria:

* people with chronic disease

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Group A Streptekok infections in rapid antigen test | Total 20 weeks
  Children with symptoms of infection will be referred to the family physician to have a rapid antigen test and to report the result to the researcher.
Incidence of symptoms of acute upper respiratory tract infection | Total 20 weeks
  Ten identified upper respiratory tract symptoms (fever, sore throat, runny nose, etc.) will be recorded weekly by family of children. The researcher will receive symptom information from the family via weekly sms
school absenteeism | Total 20 weeks
  The number of days the child does not attend school due to illness and the percentage of absenteeism

SECONDARY OUTCOMES:
Pollution rate of hands | From date of randomization until the date of first documented progression assessed up to 7 months
  Glogerm gel applied hands will shine areas containing microorganisms. Contamination rate will be calculated by taking the photo of the hands and performing brightness analysis in adobe photoshop program.

CONTACTS AND LOCATIONS:
Overall Officials: Şafak Dağhan, Study Director — Ege University, Nursing Faculty
Locations (1):
- Gülçin Uyanık, Izmir, Cigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tai JW, Mok ES, Ching PT, Seto WH, Pittet D. Nurses and physicians' perceptions of the importance and impact of healthcare-associated infections and hand hygiene: a multi-center exploratory study in Hong Kong. Infection. 2009 Aug;37(4):320-33. doi: 10.1007/s15010-009-8245-x. Epub 2009 Jul 27. PMID 19636497